CLINICAL TRIAL: NCT06930079
Title: Observational, Prospective Single-center Study on the Results of Endoscopic Injection of Autologous, Activated and Emulsified Fat in Chronic Fistulas of the Gastrointestinal Tract and Pelvic Organs
Brief Title: Endoscopic Injection of Autologous, Activated and Emulsified Fat in Chronic Fistulas of the Gastrointestinal Tract and Pelvic Organs
Acronym: ERG
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BOSKOSKI IVO, prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7097
Record Dates: First submitted 2025-03-20; First posted 2025-04-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Fistula Repair
Keywords: fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic fistulas of the GI tract or pelvic organs: Autologous activated fat tissue injection

SUMMARY:
Fistulas are defined as pathologic communications between two epithelialized surfaces and represent a complex nosologic entity that often exposes the patient to life-threatening or disabling sequelae. Their etiology can vary widely (spontaneous, iatrogenic, post-surgical perforation, anastomotic dehiscence, inflammatory process) and their treatment is complex, sometimes unresolved, and often requires a multidisciplinary approach. The chronicity of digestive and pelvic organ fistulas (e.g., vagino-vesical fistulas) is related to tissue repair mechanisms, which are delayed and subverted in favor of fibrotic and inflammatory processes. In these cases, the wound healing cascade stops at the inflammatory phase and does not result in the proliferation phase. The transition depends on changing levels of cytokines and growth factors. In the persistence of the inflammatory phase, polymorphonucleates and macrophages are active, phagocytosing and releasing enzymes that also damage healthy tissue. In this context, the anti-inflammatory, angiogenic, antiapoptotic, and tissue regenerative effects of adipose tissue-derived stromal or stem cells (ADSCs) could play a decisive role. In fact, ADSCs exhibit immunosuppressive properties on the proliferation of T cells, B lymphocytes, dendritic cells, and natural killer cells and modulate inflammation by implanting a regenerative niche with appropriate paracrine communication and subsequent tissue regeneration. "Fat grafting" has a wide range of application: it started with plastic surgery and regenerative medicine, then in orthopedics, maxillofacial surgery, and vascular surgery. Since 2019, a new procedure using processed fat grafting for the treatment of chronic fistulas of the gastrointestinal tract and pelvic organs has been initiated at the Agostino Gemelli IRCCS University Polyclinic Foundation and has become "standard of care," with good results. The procedure is quick, safe, minimally invasive and cost-effective. Subcutaneous fat, immediately after harvesting from the same patient, is mechanically stimulated with oscillatory movements, then injected under endoscopic vision directly onto the orifice of the fistula. When the fat is centrifuged, it stimulates the activation of various mesenchymal stemness-related genes, such as Sox2, Nanog and Oct4. The increase in mRNAs is tens to hundreds of times and is accompanied by a pronounced increase in the expression of the anti-inflammatory protein TSG6 and suppression of TNFalpha, normally expressed by adipose tissue.

The objective of the study is to treat chronic fistula of the gastrointestinal tract and pelvic organs of any type, symptomatic and/or impacting quality of life, in whom all other treatments (medical, endoscopic, or surgical) have failed or are not candidates.

Our primary endpoint is to evaluate the efficacy of the injection of autologous activated adipose tissue injection in these cases. Secondary endpoints evaluate the changes in patients' quality of life and the long-term efficacy of the activated fat injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients having a diagnosis of chronic fistula (diagnosis at least 3 months before the enrollment) of the pelvic organs and/or the gastrointestinal tract of any type, being symptomatic and/or impacting the quality of life.
* Age of at least 18 years.
* Able to comply with study requirements and understand and sign the Informed Consent Form.

Exclusion Criteria:

* Impaired hemostasis or any contraindication to perform endoscopy or liposuction.
* Any contraindication to perform deep sedation or general anesthesia.
* Woman being pregnant at the time of the procedure.
* Malignancy in active treatment.
* Any health issue that might put the patient at risk if the treatment is performed is judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic fistula of the pelvic organs and/or the gastrointestinal tract of any type, being symptomatic and/or impacting the quality of life
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
number of participants with fistula resolution at 6 months after the procedure. | 6 months
  Endoscopic and/or radiological evaluation

SECONDARY OUTCOMES:
number of participants with fistula resolution at 2 months after the procedure. | 2 months
  Endoscopic evaluation
Quality of life measure before and after the procedure | 12 months
  Short Form Health Survey 36 (SF-36) test will be administered at screening visit, then at 6 and 12 months after the procedure; 0 is the worst possible outcome and 100 is the best possible outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No